CLINICAL TRIAL: NCT04089215
Title: A Phase II Open-Label, Single-Arm, Multicenter Study of JWCAR029, CD19-targeted Chimeric Antigen Receptor (CAR) T Cells for Relapsed and Refractory (R/R) Non-Hodgkins Lymphoma
Brief Title: CD19-targeted CAR T Cells for Relapsed and Refractory (R/R) Non-Hodgkins Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029-002
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma, Non-Hodgkin; Diffuse Large B Cell Lymphoma; Follicular Lymphoma
Keywords: JWCAR029; B-Cell Malignancies; non-Hodgkin lymphoma; CAR T cells; Chimeric antigen receptor; Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Recurrence | interventions — Automobiles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR029 treatment (Experimental): JWCAR029 be administrated in two dose level
  Interventions: Biological: CD19-targeted Chimeric Antigen Receptor (CAR) T Cells

INTERVENTIONS:
Biological: CD19-targeted Chimeric Antigen Receptor (CAR) T Cells — JWCAR029 be administered at dose level: 1 x 10^8 CAR+T cells and 1.5 x 10^8 CAR+T cells

SUMMARY:
This is a phase II, open-label, single-arm, multicenter study to asess the efficacy and safety of JWCAR029 in adult R/R Non-Hodgkins Lymphoma subjects in China.

DETAILED DESCRIPTION:
This is a phase II, open-label, single-arm, multicenter study conducted in adult subjects with R/R Non-Hodgkins Lymphoma in China to evaluate the safety, efficacy, pharmacokinetics(PK), pharmacodynamics(PD) of JWCAR029 and collect the patient reported quality of life changes and immune response after JWCAR029 treatment.

There will be two cohorts of cohort A and cohort B. Large B cell lymphoma (LBCL) patients will be enrolled in cohort A and follicular lymphoma patients will be enrolled in cohort B. Two dose levels of 1.0 x 10^8 CAR+ T cells and 1.5 x 10^8 CAR+ T cells are adopted in this study in both cohorts, subjects will be randomly assigned into the two dose levels with a 1:1 ratio. All sujects will be followed for 2 years following JWCAR029 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to participate in the study:

  1. ≥ 18 years old;
  2. Sign on the informed consent;
  3. Subject must have histologically confirmed large B lymphoma or follicular lymphoma;
  4. Subjects have accessible PET-positive lesion and have measurable CT-positive lesion according to Lugano Classification;
  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
  6. Adequate organ function;
  7. Adequate vascular access for leukapheresis procedure;
  8. Subjects who have previously received CD19 targeted therapy must confirm that lymphoma lesions still express CD19;
  9. Women of childbearing potential must agree to use highly effective methods of contraception for 1 year after the last dose of JWCAR029;
  10. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 1 year after the last dose of JWCAR029.

Exclusion Criteria:

1. Central nervous system (CNS) only involvement by malignancy or primary CNS lymphoma;
2. History of another primary malignancy that has not been in remission for at least 2 years;
3. Subjects has HBV, HCV, HIV or syphilis infection at the time of screening;
4. Deep venous thrombosis (DVT)/Pulmonary embolism (PE), or DVT/PE requires anti-coagulation within 3 months prior to signing the ICF;
5. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection;
6. Presence of acute or chronic graft-versus-host disease (GVHD);
7. History of any serious cardiovascular disease or presence of clinically relevant CNS pathology;
8. Pregnant or nursing women;
9. Subjects using of any chemotherapy, corticisteriod, experiment agents, GVHD therapies, radiation, allo-HSCT or any other therapies for lymphoma must go through a specific wash-out period before leukapheresis;
10. Uncontrolled conditions or unwillingness or inability to follow the procedures required in the protocol;
11. Received CAR T-cell or other genetically-modified T-cell therapy previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) in LBCL subjects in cohort A; | 3 months
  Objective response rate (ORR) in 3 month in cohort A of large B cell lymphoma (LBCL) subjects；
Complete response rate (CRR) in FL subjects in cohort B | 3 months
  Complete response rate (CRR) in 3 month in cohort B of follicular lymphoma (FL) subjects

SECONDARY OUTCOMES:
Complete response rate (CRR) in cohort A of LBCL subjects | 3 months
Objective response rate (ORR) in cohort B of FL subjects | 3 months
Adverse events (AEs) | up to 24 months after JWCAR029 infusion
  Number of participants with adverse events, type of adverse events, severity of adverse events, and number of participants with laboratory abnormalities, type of laboratory abnormalities and severity of laboratory abnormalities.
Duration of response (DOR) | up to 24 months after JWCAR029 infusion
  Time from first response(PR or CR) to disease progression or death from any cause.
Duration of complete remission (DoCR) | up to 24 months after JWCAR029 infusion
  Time from complete response (CR) to disease progression or death from any cause.
Duration of partial remission (DoPR) | up to 24 months after JWCAR029 infusion
  Time from partial response (PR) to disease progression or death from any cause.
Time to response (TTR) | up to 24 months after JWCAR029 infusion
  Time from JWCAR029 infusion to first documentation of CR or PR
Time to complete response (TTCR) | up to 24 months after JWCAR029 infusion
  Time from JWCAR029 infusion to first documentation of CR
Pharmacokinetic (PK)- Cmax of JWCAR029 | up to 1 year after JWCAR029 infusion
  Maximum observed concentration of JWCAR029 in peripheral blood
Pharmacokinetic (PK)- Tmax of JWCAR029 | up to 1 year after JWCAR029 infusion
  Time to maximum concentration of JWCAR029 in the peripheral blood
Pharmacokinetic (PK)- AUC of JWCAR029 | up to 1 year after JWCAR029 infusion
  Area under the concentration vs time curve of JWCAR029
Progression-free survival (PFS) | 3 to 5 years after JWCAR029 infusion
Overall survival | 3 to 5 years after JWCAR029 infusion
Quality of Life C30 questionnaire (EORTC-QLQ-C30) | up to 2 year after JWCAR029 infusion
  EORTC-QLQ-C30 is composed of both multi-item scales and single item measures. These include five functional scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, nausea/vomiting, and pain), a global health status/health-related quality of life (HRQoL) scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Each of the multi-item scales includes a different set of items - no item occurs in more than one scale
European Quality of Life-5 Dimensions health state classifier to 5 Levels (EQ-5D-5L) | up to 2 year after JWCAR029 infusion
  The EQ-5D-5L consists of the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems)
ICU and non-ICU hospitalization days | up to 2 year after JWCAR029 infusion
ICU and non-ICU hospitalization reasons | up to 2 year after JWCAR029 infusion
Anti-therapeutic JWCAR029 antibody | up to 2 year after JWCAR029 infusion
Changes of T cell counts, subgroups and serum cytokines | up to 2 year after JWCAR029 infusion
CD19 expression in tumor biopsy samples | up to 2 year after JWCAR029 infusion
Changes of inflammation biomarkers-CRP | up to 1 year after JWCAR029 infusion
Changes of inflammation biomarkers-serum ferritin | up to 1 year after JWCAR029 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (10):
- China (10):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhenzhou Universtity, Zhenzhou, Henan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Institute of Hematology&Hospital of Blood Disease CAMS, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ying Z, Yang H, Guo Y, Li W, Zou D, Zhou D, Wang Z, Zhang M, Wu J, Liu H, Zhang P, Yang S, Zhou Z, Zheng H, Song Y, Zhu J. Relmacabtagene autoleucel (relma-cel) CD19 CAR-T therapy for adults with heavily pretreated relapsed/refractory large B-cell lymphoma in China. Cancer Med. 2021 Feb;10(3):999-1011. doi: 10.1002/cam4.3686. Epub 2020 Dec 31. PMID 33382529
- [Derived] Song Y, Zou D, Yang H, Wu J, Guo Y, Li W, Liu H, Xia Z, Zhang Y, Zhou Z, Zhu J. Two-year follow-up of relmacabtagene autoleucel in relapsed or refractory follicular lymphoma in RELIANCE study. Br J Haematol. 2025 Oct;207(4):1476-1483. doi: 10.1111/bjh.20122. Epub 2025 Sep 1. PMID 40888120
- [Derived] Ying Z, Yang H, Guo Y, Li W, Zou D, Zhou D, Wang Z, Zhang M, Wu J, Liu H, Wang C, Ma L, Yang S, Zhou Z, Qin Y, Song Y, Zhu J. Long-term outcomes of relmacabtagene autoleucel in Chinese patients with relapsed/refractory large B-cell lymphoma: Updated results of the RELIANCE study. Cytotherapy. 2023 May;25(5):521-529. doi: 10.1016/j.jcyt.2022.10.011. Epub 2023 Feb 24. PMID 36842849
- [Derived] Ying Z, Zou D, Yang H, Wu J, Guo Y, Li W, Liu H, Wang C, Ma L, Yang S, Zhou Z, Qin Y, Song Y, Zhu J. Preliminary efficacy and safety of Relmacabtagene autoleucel (Carteyva) in adults with relapsed/refractory follicular lymphoma in China: A phase I/II clinical trial. Am J Hematol. 2022 Dec;97(12):E436-E438. doi: 10.1002/ajh.26711. Epub 2022 Sep 14. No abstract available. PMID 36053875